CLINICAL TRIAL: NCT02316444
Title: Strategies for the Prevention of Hepatitis B Viral Infection Among HIV Infected Adults in Uganda
Brief Title: Strategies for the Prevention of Hepatitis B Among HIV Infected Patients in Uganda
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Makerere University (Other); Uganda Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: U010
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: HIV/AIDS and Infections
Keywords: Hepatitis B vaccine HIV infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — Hepatitis B Vaccines; Euvax-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAART exposed (Other): Participants in both arms will receive the Hepatitis B vaccine as summarized in the study description
  Interventions: Biological: Hepatitis B vaccine
- HAART naive (Other): Participants in both arms will receive the Hepatitis B vaccine as summarized in the study description
  Interventions: Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: Hepatitis B vaccine — An eligible participant will receive 3 doses of hepatitis B vaccine ( 20mcg in the deltoid intramuscular). Then their immune response will be assessed. Non responders will receive 3 additional vaccine doses off protocol
  Other Names: Euvax B (Sonafi)

SUMMARY:
The aim of this study is to compare the effectiveness of two vaccination strategies against Hepatitis B virus (HBV) in subjects already infected with human immunodeficiency virus (HIV).

Researchers plan to determine the optimal vaccination strategy for achieving protective immunity to HBV infection in HIV-infected adults attending Mulago Hospital's HIV care clinic.

Primary objectives are to assess:

1. The role of CD4-cell count and HIV viral loads on the HBV vaccine response.
2. The role of highly active antiretroviral therapy (HAART) on the HBV vaccine response.

The secondary objective is to evaluate whether lack of HAART is associated with high rates of loss to follow-up.

DETAILED DESCRIPTION:
This is an interventional study in which researchers will recruit HIV positive individuals who do not have hepatitis B (HBV negative) in order to assess the effectiveness of a hepatitis B vaccine in 2 subgroups:

1. Those who have received less than 3 months treatment, or no treatment, with highly active antiretroviral drugs (HAART naive).
2. Those who have received at least 3 months of treatment with highly active antiretroviral drugs (HAART exposed).

All study participants will receive vaccination against HBV.

There will be 6-12 clinic visits depending on 1) whether or not the participant responds to the standard 3-dose vaccination protocol and 2) whether he or she suffers a clinical condition or vaccine related adverse event that would call for postponement of the next vaccine dose.

The first visit will be to determine if the participant is eligible for the study. If eligible, the participant will receive one dose of vaccine at each of the following three visits. The fifth visit will be to collect blood to determine whether the participant has responded to the 3-dose vaccination protocol. The sixth visit will be to discuss the outcome of the vaccination with the participant. Participants who respond favorably to the 3-dose vaccine protocol will exit the study at this point. However, if a participant fails to respond to the initial 3-dose vaccine protocol, he or she may restart the regimen and receive another 3 doses of vaccine following the same schedule as before but off protocol.

Participants will be reimbursed for travel costs to and from the clinic for scheduled clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatitis B core antibody (anti-HBc) and anti-HBs negative
2. Age ≥18 years
3. HIV infected persons (HAART naïve and HAART exposed). HAART enrollees will be considered to be HAART exposed if they have been taking these medications for at least 3 months. Participants that have never been on HAART and those that have been on HAART for <3months will be considered to be HAART naïve. HAART exposed enrollees will have an adherence of at least 95%.
4. Ambulatory
5. Intention to attend the Mulago HIV/AIDS clinic for the 18 months
6. Able and willing to comply with study protocol including providing informed consent

Exclusion Criteria:

1. History of hypersensitivity to vaccines or intolerance to any of the HBV vaccine components
2. Previously-confirmed diagnosis of decompensated liver disease or HCC
3. Serological evidence of prior receipt of the HBV vaccine (anti-HBS positive, anti-HBc negative) or documented (clinical) evidence of having been vaccinated.
4. Known history of HBV infection (HBsAg and/or anti-HBc positive).
5. Inability to follow study procedures
6. If a participant chooses not to consent to the review of his or her medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Hepatitis B virus (HBV) vaccine response | 18 months
  Measure Hepatitis B surface antibody (anti-HBs) levels and cell mediated immune response.

SECONDARY OUTCOMES:
Loss to follow-up (HAART naive vs. HAART exposed individuals) | 18 months
  Compare the number of individuals lost to follow-up among the HAART naive and HAART exposed.

CONTACTS AND LOCATIONS:
Overall Officials: Ponsiano Ocama, PhD, Principal Investigator — Makerere University; Corey Casper, MD, Principal Investigator — Fred Hutchinson Cancer Center; Emmanuel Seremba, MMED, Principal Investigator — HCRI-Ug, Makerere University
Locations (1):
- Mulago National referral hospital, Kampala, Uganda